CLINICAL TRIAL: NCT04751591
Title: Prospective Randomized Controlled Multicenter Clinical Trial For Comparison Of Safety Between Endoscopic Resection And Laparoscopic Partial Gastrectomy In Patients With 2-5cm Gastric Gastrointestinal Stromal Tumor
Brief Title: Study On Safety Of Endoscopic Resection For 2-5cm Gastric Gastrointestinal Stromal Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SK2020-032
Record Dates: First submitted 2021-01-30; First posted 2021-02-12 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Gastric GIST
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic resection (Experimental): The endoscopist will perform endoscopic resection for patients enrolled in this group.
  Interventions: Procedure: Endoscopic resection
- Laparoscopic partial gastrectomy (Other): The endoscopist will perform laparoscopic partial gastrectomy for patients enrolled in this group.
  Interventions: Procedure: Laparoscopic partial gastrectomy

INTERVENTIONS:
Procedure: Endoscopic resection — Endoscopic submucosal dissection (ESD) or endoscopic full-thickness resection (EFTR) for patients with 2-5cm gastric GISTs
  Arms: Endoscopic resection
Procedure: Laparoscopic partial gastrectomy — Laparoscopic partial gastrectomy for patients with 2-5cm gastric GISTs
  Arms: Laparoscopic partial gastrectomy

SUMMARY:
This research is a prospective, multi-center trial for endoscopic resection and laparoscopic partial gastrectomy in patients with 2-5cm gastric gastrointestinal stromal tumor. The primary purpose of this study is to evaluate the early operative morbidity and mortality and determine the safety of endoscopic resection compared with laparoscopic partial gastrectomy for 2-5cm gastric gastrointestinal stromal tumor. The second purpose is to evaluate the recovery course and compare the postoperative hospital stay of the patients enrolled in this study.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors (GIST) originate from interstitial cells of Cajal (ICC) and are the most common tumors derived from mesenchymal tissues of the digestive tract. GISTs can occur in any part of the digestive tract, among which gastric stromal tumors are the most common, accounting for about 60%. The incidence of GIST has been increasing in recent years, partly due to the gradual popularity of gastrointestinal endoscopy. Many early GISTs with smaller tumors have also received early diagnosis and treatment intervention. Due to the potential malignancy of GISTs, complete resection of the tumor is the first and only radical treatment option currently.

Many studies have shown that laparoscopy is safe and effective approach in the treatment of gastric stromal tumors. In principle, as long as the tumor can be completely resected (neither residue macro nor microscopic) with intact tumor capsule and without tumor rupture, laparoscopic surgery is definite an option. Studies showed both short-term and long-term results of laparoscopic surgery were comparable to conventional open surgeries.

On the other hand, endoscopic resection showed promising results in recent years. Endoscopic submucosal dissection endoscopic full-thickness resection are both reported with promising results in terms of safety and short-term efficacy.

Though endoscopic resection has been suggested as one of the treatment options for gastric GISTs, No randomized controlled trial for endoscopic resection versus laparoscopic partial gastrectomy exists at this moment. This research is a prospective, multi-center trial for endoscopic resection and laparoscopic partial gastrectomy in patients with 2-5cm gastric GISTs. The primary purpose of this study is to evaluate the early operative morbidity and mortality and determine the safety of endoscopic resection compared with laparoscopic partial gastrectomy for 2-5cm gastric GISTs. The second purpose is to evaluate the recovery course and compare the postoperative hospital stay of the patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gastric GISTs in imaging examinations including contrast-enhanced abdominal and pelvic CT, EGD examination and endoscopic ultrasound examination
* The maximum diameter of the tumor is > 2cm and ≤ 5cm
* No history of upper abdominal surgery (except for laparoscopic cholecystectomy)
* No history of neoadjuvant therapy or targeted therapy
* Preoperative performance status (ECOG，Eastern Cooperative Oncology Group) of 0 or 1
* Preoperative ASA (American Society of Anesthesiologists) scoring: I-III
* Sufficient organ functions
* Written informed consent

Exclusion Criteria:

* Gastric GISTs with completely extra-luminal growth pattern
* Metastases found in preopreative examinations
* History of simultaneous malignancies or heterochronous malignancies within 5 years
* Women during pregnancy or breast-feeding
* Severe heart and lung disease, severe renal insufficiency, unable to perform laparoscopic surgery
* Body temperature ≥ 38℃ before surgery or infectious disease with a systemic therapy indicated
* Severe mental disease
* Severe respiratory disease
* Severe hepatic and renal dysfunction
* Unstable angina pectoris or history of myocardial infarction within 6 months
* History of cerebral infarction or cerebral hemorrhage within 6 months
* Patients with other diseases who can be surgically intervened at the same time
* Continuous systemic steroid therapy within 1 month (except for topical use)
* Patients are participating or have participated in another clinical trial (within 6 months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Early operative morbidity rate | 30 days
  The early operative morbidity is defined as the event observed within 30 days following surgery, including intraoperative and postoperative complications.
Early operative mortality rate | 30 days
  The early operative mortality is defined as deaths observed within 30 days following surgery.

SECONDARY OUTCOMES:
Operation time | intraoperative
  Operation time is documented as a composite outcome measure.
Time to first ambulation | 30 days
  Time to first ambulation is used to assess the postoperative recovery course, which is a composite outcome measure.
Time to first flatus | 30 days
  Time to first flatus is used to assess the postoperative recovery course, which is a composite outcome measure.
Time to first liquid diet | 30 days
  Time to first liquid diet is used to assess the postoperative recovery course, which is a composite outcome measure.
Time to first soft diet | 30 days
  Time to first soft diet is used to assess the postoperative recovery course, which is a composite outcome measure.
Postoperative hospital stay | 30 days
  The length of postoperative hospital stay will be recorded.
En bloc resection rate | 0, day of endoscopic surgery or laparoscopic surgery
  The rate of en bloc resection in all cases will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Pinghong Zhou, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon JG, Hwang SJ, Hennig GW, Bayguinov Y, McCann C, Chen H, Rossi F, Besmer P, Sanders KM, Ward SM. Changes in the structure and function of ICC networks in ICC hyperplasia and gastrointestinal stromal tumors. Gastroenterology. 2009 Feb;136(2):630-9. doi: 10.1053/j.gastro.2008.10.031. Epub 2008 Nov 1. PMID 19032955
- [Background] Heinrich MC, Rubin BP, Longley BJ, Fletcher JA. Biology and genetic aspects of gastrointestinal stromal tumors: KIT activation and cytogenetic alterations. Hum Pathol. 2002 May;33(5):484-95. doi: 10.1053/hupa.2002.124124. PMID 12094373
- [Background] Bamboat ZM, Dematteo RP. Updates on the management of gastrointestinal stromal tumors. Surg Oncol Clin N Am. 2012 Apr;21(2):301-16. doi: 10.1016/j.soc.2011.12.004. PMID 22365521
- [Background] Steigen SE, Eide TJ. Trends in incidence and survival of mesenchymal neoplasm of the digestive tract within a defined population of northern Norway. APMIS. 2006 Mar;114(3):192-200. doi: 10.1111/j.1600-0463.2006.apm_261.x. PMID 16643186
- [Background] Demetri GD, von Mehren M, Antonescu CR, DeMatteo RP, Ganjoo KN, Maki RG, Pisters PW, Raut CP, Riedel RF, Schuetze S, Sundar HM, Trent JC, Wayne JD. NCCN Task Force report: update on the management of patients with gastrointestinal stromal tumors. J Natl Compr Canc Netw. 2010 Apr;8 Suppl 2(0 2):S1-41; quiz S42-4. doi: 10.6004/jnccn.2010.0116. PMID 20457867
- [Background] Pucci MJ, Berger AC, Lim PW, Chojnacki KA, Rosato EL, Palazzo F. Laparoscopic approaches to gastric gastrointestinal stromal tumors: an institutional review of 57 cases. Surg Endosc. 2012 Dec;26(12):3509-14. doi: 10.1007/s00464-012-2374-5. Epub 2012 Jun 9. PMID 22684977
- [Background] Ohtani H, Maeda K, Noda E, Nagahara H, Shibutani M, Ohira M, Muguruma K, Tanaka H, Kubo N, Toyokawa T, Sakurai K, Yamashita Y, Yamamoto A, Hirakawa K. Meta-analysis of laparoscopic and open surgery for gastric gastrointestinal stromal tumor. Anticancer Res. 2013 Nov;33(11):5031-41. PMID 24222147
- [Background] He Z, Sun C, Zheng Z, Yu Q, Wang T, Chen X, Cao H, Liu W, Wang B. Endoscopic submucosal dissection of large gastrointestinal stromal tumors in the esophagus and stomach. J Gastroenterol Hepatol. 2013 Feb;28(2):262-7. doi: 10.1111/jgh.12056. PMID 23190047
- [Background] Zhou PH, Yao LQ, Qin XY, Cai MY, Xu MD, Zhong YS, Chen WF, Zhang YQ, Qin WZ, Hu JW, Liu JZ. Endoscopic full-thickness resection without laparoscopic assistance for gastric submucosal tumors originated from the muscularis propria. Surg Endosc. 2011 Sep;25(9):2926-31. doi: 10.1007/s00464-011-1644-y. Epub 2011 Mar 18. PMID 21424195
- [Background] Chen T, Zhou PH, Chu Y, Zhang YQ, Chen WF, Ji Y, Yao LQ, Xu MD. Long-term Outcomes of Submucosal Tunneling Endoscopic Resection for Upper Gastrointestinal Submucosal Tumors. Ann Surg. 2017 Feb;265(2):363-369. doi: 10.1097/SLA.0000000000001650. PMID 28059965
- [Background] ASGE Technology Committee; Aslanian HR, Sethi A, Bhutani MS, Goodman AJ, Krishnan K, Lichtenstein DR, Melson J, Navaneethan U, Pannala R, Parsi MA, Schulman AR, Sullivan SA, Thosani N, Trikudanathan G, Trindade AJ, Watson RR, Maple JT. ASGE guideline for endoscopic full-thickness resection and submucosal tunnel endoscopic resection. VideoGIE. 2019 Jun 29;4(8):343-350. doi: 10.1016/j.vgie.2019.03.010. eCollection 2019 Aug. PMID 31388606
- [Background] Wang C, Gao Z, Shen K, Cao J, Shen Z, Jiang K, Wang S, Ye Y. Safety and efficiency of endoscopic resection versus laparoscopic resection in gastric gastrointestinal stromal tumours: A systematic review and meta-analysis. Eur J Surg Oncol. 2020 Apr;46(4 Pt A):667-674. doi: 10.1016/j.ejso.2019.10.030. Epub 2019 Dec 13. PMID 31864827
- [Background] Wang H, Feng X, Ye S, Wang J, Liang J, Mai S, Lai M, Feng H, Wang G, Zhou Y. A comparison of the efficacy and safety of endoscopic full-thickness resection and laparoscopic-assisted surgery for small gastrointestinal stromal tumors. Surg Endosc. 2016 Aug;30(8):3357-61. doi: 10.1007/s00464-015-4612-0. Epub 2015 Oct 23. PMID 26497947
- [Background] Yin X, Yin Y, Chen H, Shen C, Tang S, Cai Z, Zhang B, Chen Z. Comparison Analysis of Three Different Types of Minimally Invasive Procedures for Gastrointestinal Stromal Tumors </=5 cm. J Laparoendosc Adv Surg Tech A. 2018 Jan;28(1):58-64. doi: 10.1089/lap.2017.0305. Epub 2017 Oct 30. PMID 29083255
- [Background] Wu CR, Huang LY, Guo J, Zhang B, Cui J, Sun CM, Jiang LX, Wang ZH, Ju AH. Clinical Control Study of Endoscopic Full-thickness Resection and Laparoscopic Surgery in the Treatment of Gastric Tumors Arising from the Muscularis Propria. Chin Med J (Engl). 2015 Jun 5;128(11):1455-9. doi: 10.4103/0366-6999.157651. PMID 26021500
- [Background] Huang LY, Cui J, Wu CR, Zhang B, Jiang LX, Xian XS, Lin SJ, Xu N, Cao XL, Wang ZH. Endoscopic full-thickness resection and laparoscopic surgery for treatment of gastric stromal tumors. World J Gastroenterol. 2014 Jul 7;20(25):8253-9. doi: 10.3748/wjg.v20.i25.8253. PMID 25009400
- [Background] Chen L, Zhang Q, Li FY, Yang L, Zhang DC, Wang LJ, Wang WZ, Li Z, Xu JH, He ZY, Xu KJ, Chen M, Xu H, Xu ZK. Comparison of treatment outcomes between laparoscopic and endoscopic surgeries for relatively small gastric gastrointestinal stromal tumors. Surg Oncol. 2018 Dec;27(4):737-742. doi: 10.1016/j.suronc.2018.10.002. Epub 2018 Oct 2. PMID 30449501
- [Background] Zhao Y, Pang T, Zhang B, Wang L, Lv Y, Ling T, Zhang X, Huang Q, Xu G, Zou X. Retrospective Comparison of Endoscopic Full-Thickness Versus Laparoscopic or Surgical Resection of Small (</= 5 cm) Gastric Gastrointestinal Stromal Tumors. J Gastrointest Surg. 2020 Dec;24(12):2714-2721. doi: 10.1007/s11605-019-04493-6. Epub 2019 Dec 10. PMID 31823317